CLINICAL TRIAL: NCT05676931
Title: A Phase II, Open-label, Platform Study, to Evaluate Immunotherapy-based Combinations in Participants With Advanced Non-Small Cell Lung Cancer
Brief Title: Study With Various Immunotherapy Treatments in Participants With Lung Cancer
Acronym: EDGE-Lung
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EDGE-Lung; 2022-502916-35-01 (EU CTIS Number)
Record Dates: First submitted 2022-12-09; First posted 2023-01-09 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Advanced Non-Small Cell Lung Cancer
Keywords: Advanced Non-Small Cell Lung Cancer; Domvanalimab; Zimberelimab; Quemliclustat; Anti-TIGIT antibody; Anti-PD-1 antibody
MeSH Terms: interventions — quemliclustat; zimberelimab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- A1: Domvanalimab + Zimberelimab (Experimental): Domvanalimab and Zimberelimab, both administered by IV infusion
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab
- A2: Domvanalimab + Zimberelimab (Experimental): Domvanalimab and Zimberelimab, both administered by IV infusion
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab
- A3: Quemliclustat + Zimberelimab (Experimental): Quemliclustat and Zimberelimab, both administered by IV infusion
  Interventions: Drug: Quemliclustat; Drug: Zimberelimab
- B1: Quemliclustat + Zimberelimab + Platinum Doublet Chemotherapy (Experimental): Quemliclustat, zimberelimab, and platinum doublet chemotherapy, all administered by IV infusion
  Interventions: Drug: Quemliclustat; Drug: Zimberelimab; Drug: Platinum-Based Doublet
- B2: Domvanalimab + Zimberelimab + Platinum Doublet Chemotherapy (Experimental): Domvanalimab, Zimberelimab, and platinum doublet chemotherapy, all administered by IV infusion
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab; Drug: Platinum-Based Doublet
- B3: Domvanalimab + Quemliclustat + Zimberelimab + Platinum Doublet Chemotherapy (Experimental): Domvanalimab, Quemliclustat, Zimberelimab, and platinum doublet chemotherapy, all administered by IV infusion
  Interventions: Drug: Domvanalimab; Drug: Quemliclustat; Drug: Zimberelimab; Drug: Platinum-Based Doublet
- B4: Domvanalimab + Zimberelimab + Platinum Doublet Chemotherapy (Experimental): Domvanalimab, Zimberelimab, and platinum doublet chemotherapy, all administered by IV infusion
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab; Drug: Platinum-Based Doublet
- B5: Domvanalimab + Zimberelimab + Platinum Doublet Chemotherapy (Experimental): Domvanalimab, Zimberelimab, and platinum doublet chemotherapy, all administered by IV infusion
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab; Drug: Platinum-Based Doublet
- C1: Quemliclustat + Zimberelimab + Docetaxel (Experimental): Quemliclustat, Zimberelimab, and Docetaxel, all administered by IV infusion
  Interventions: Drug: Quemliclustat; Drug: Zimberelimab; Drug: Docetaxel
- C2: Domvanalimab + Zimberelimab + Docetaxel (Experimental): Domvanalimab, Zimberelimab, and Docetaxel, all administered by IV infusion
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab; Drug: Docetaxel

INTERVENTIONS:
Drug: Domvanalimab — Administered as specified in the treatment arm
  Arms: A1: Domvanalimab + Zimberelimab; A2: Domvanalimab + Zimberelimab; B2: Domvanalimab + Zimberelimab + Platinum Doublet Chemotherapy; B3: Domvanalimab + Quemliclustat + Zimberelimab + Platinum Doublet Chemotherapy; B4: Domvanalimab + Zimberelimab + Platinum Doublet Chemotherapy; B5: Domvanalimab + Zimberelimab + Platinum Doublet Chemotherapy; C2: Domvanalimab + Zimberelimab + Docetaxel
Drug: Quemliclustat — Administered as specified in the treatment arm
  Arms: A3: Quemliclustat + Zimberelimab; B1: Quemliclustat + Zimberelimab + Platinum Doublet Chemotherapy; B3: Domvanalimab + Quemliclustat + Zimberelimab + Platinum Doublet Chemotherapy; C1: Quemliclustat + Zimberelimab + Docetaxel
Drug: Zimberelimab — Administered as specified in the treatment arm
Drug: Docetaxel — Administered as specified in the treatment arm
  Arms: C1: Quemliclustat + Zimberelimab + Docetaxel; C2: Domvanalimab + Zimberelimab + Docetaxel
Drug: Platinum-Based Doublet — Administered as specified in the treatment arm
  Arms: B1: Quemliclustat + Zimberelimab + Platinum Doublet Chemotherapy; B2: Domvanalimab + Zimberelimab + Platinum Doublet Chemotherapy; B3: Domvanalimab + Quemliclustat + Zimberelimab + Platinum Doublet Chemotherapy; B4: Domvanalimab + Zimberelimab + Platinum Doublet Chemotherapy; B5: Domvanalimab + Zimberelimab + Platinum Doublet Chemotherapy

SUMMARY:
The purpose of this study is to assess the objective response rate (ORR) of immunotherapy-based combination therapy and to assess the safety and tolerability of immunotherapy-based combination therapy.

DETAILED DESCRIPTION:
The study includes multiple substudy arms (Substudy A, B, C), which will evaluate immunotherapy-based combinations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented Stage IV metastatic, NSCLC
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 1
* At least one measurable target lesion per RECIST v1.1.
* Adequate organ function
* Participants must be willing to provide adequate tumor tissue

Exclusion Criteria:

* Underlying medical conditions that, in the Investigator's or Sponsor's opinion, will make the administration of Investigational Product(s) (IPs) hazardous
* Use of any live vaccines against infectious diseases within 28 days of first dose of IP(s).
* Use of supra-physiologic doses of corticosteroids (> 10 mg/day of oral prednisone or equivalent) or immunosuppressive medications ≤ 14 days before the initiation of study treatment (absorbable topical corticosteroids are not excluded).
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Any active autoimmune disease or a documented history of autoimmune disease or syndrome that required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs), except for vitiligo or resolved childhood asthma/atopy

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) as measured by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | Up to 58 months
The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Up to 58 months

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of first dose until the date of death due to any cause (approximately 58 months)
Progression-free Survival (PFS) as determined by the Investigator according to RECIST v1.1 | Up to 58 months
Disease Control Rate (DCR) | Up to 58 months
Duration of response (DoR) as determined by the Investigator according to RECIST v1.1 | Up to 58 months
Investigational study treatments peak plasma or serum concentration (Cmax) | Up to 58 months
Investigational study treatments time of peak concentration (Tmax) | Up to 58 months
Investigational study treatments area under the plasma or serum concentration versus time curve (AUC) | Up to 58 months
Percentage of biologic treatment-emergent antidrug-antibody (ADA)-positive participants and ADA-negative participants | Up to 58 months

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (51):
- United States (9):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - University of California San Diego (UCSD), La Jolla, California
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Hematology Oncology Associates Of The Treasure Coast, Port Saint Lucie, Florida
  - Florida Cancer Specialists (Administration and Drug Shipment), The Villages, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Ochsner Clinic Foundation, Jefferson, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Medical Oncology Associated, PS (dba Summit Cancer Centers), Spokane, Washington
- Australia (4):
  - The Border Cancer Hospital, Albury, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Cancer Research SA Pty Ltd, Adelaide, South Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- France (4):
  - CHU Bordeaux Centre Francois Magendie Hôpital du Haut Lévèque, Bordeaux
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud, Lyon
  - Institut De Cancerologie Strasbourg Europe ICANS, Strasboug
  - Hopital FOCH, Suresnes
- Georgia (5):
  - LTD High Technology Hospital Medcenter, Batumi
  - Caucasus Medical Center, Tbilisi
  - Israel Georgian Medical Research Clinic Healthycore, Tbilisi
  - JSC K. Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - Ltd Pineo Medical Ecosystem, Tbilisi
- Italy (5):
  - Istituto Romagnolo per lo Studio dei Tumori-Dino Amadori - IRST, Meldola
  - stituto Nazionale per lo Studio e la Cura dei Tumori, Milan
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Sanitaria Territoriale Pesaro Urbino (AST PU), Pesaro
  - Fondazione IRCCS Istituto Nazionale dei tumori di Milano, Rome
- Poland (4):
  - Szpitale Pomorskie sp. z o.o, Gdynia
  - Uniwersyteckie Centrum Kliniczne, im. prof. K. Gibińskiego, Katowice
  - Medpolonia Sp. Z.o.o., Poznan
  - Centrum Onkologii - Instytut im. Marii Sk?odowskiej-Curie, Warsaw
- South Korea (5):
  - Samsung Changwon Hospital, Changwon-Si
  - Chungbuk National University Hospital, Cheongju-si
  - Chonam National University Hwasun Hospital, Hwasun-gun
  - Korea University Guro Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (10):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Mutua Terrassa, Barcelona
  - UOMI Cancer Centre, Barcelona
  - Complejo Hospitalario Universitario Insular Materno Infantil De Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Quirónsalud Málaga, Málaga
  - Hospital Universitario De La Virgen De Valme, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital 9 de Octubre Vithas Valencia, Valencia
  - Hospital Universitario y Politécnico la Fe, Valencia
- Taiwan (4):
  - E-DA Healthcare Group E-DA Hospital, Kaoshiung
  - Taipei Medical University - Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - Mackey Memorial Hospital, Taipei
  - National Taiwan University Hospital Yumlin Branch, Yunlin County
- Barts Health NHS Trust St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No